CLINICAL TRIAL: NCT06059976
Title: EVALUATION OF PRACTICES: RETROSPECTIVE AND PROSPECTIVE MONOCENTRIC SURVEY ON THE SATISFACTION OF PATIENTS UNDERGOING CARDIAC SURGERY WHO WERE ABLE TO BENEFIT FROM ADDITIONAL MANAGEMENT BY ERICKSONIAN MEDICAL HYPNOSIS DURING THEIR STAY
Brief Title: HYPNOSIS DURING PERIOPERATIVE CARDIAC SURGERY
Acronym: OCEANIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00916-39
Record Dates: First submitted 2023-09-19; First posted 2023-09-29 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Hypnosis With Cardiac Surgery
Keywords: hypnosis; cardiac surgery; peri operatoire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypnosis: Inclusion of patients undergoing major cardiac surgery who have received perioperative hypnosis sessions from January 2023.
  After obtaining their consent to participate in this study

SUMMARY:
Evaluation of practices: retrospective and prospective monocentric survey on the satisfaction of patients undergoing Cardiac Surgery who were able to benefit from additional management by Ericksonian Medical Hypnosis during their stay.

DETAILED DESCRIPTION:
Since 2018, additional care using Ericksonian Medical Hypnosis has been offered to patients undergoing cardiac surgery. Cardiac surgery is one of the most complex and high-risk procedures, requiring a general anaesthetic and a stay in intensive care.

Its aim is to reduce pre-operative stress and anxiety, which are always present to varying degrees before this type of treatment. The aim is to put the patient back at the centre of his or her care by making them active and active participants throughout the treatment process.

Many studies have demonstrated the benefits of hypnosis in reducing anxiety, depression, pain perception, sedation and comfort during hospitalisation. However, very few studies have looked at the quality of life of these patients for up to a year.

Hypnosis support is subject to the number and presence of trained nursing staff.

In order to assess the feelings of patients who have benefited from this additional treatment, and to improve our practices, we would like to carry out a satisfaction survey using questionnaires including the EQ5D-5L quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Patients undergoing major cardiac surgery
* Patients who have had perioperative hypnosis sessions.

Exclusion Criteria:

* Opposition of the patient to the conservation of data
* Subject under guardianship or subject deprived of liberty, as referred to in articles L1121-5 to L1121-8 of the CSP (French Public Health Code)
* Pregnant or breast-feeding women
* Contraindication to the practice of hypnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalised for cardiac surgery who received hypnosis sessions in cardiac surgery at their request.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feelings of patients who received perioperative support using Ericksonian hypnosis during their cardiac surgery treatment. | 1 years
  Perioperative Ericksonian hypnosis satisfaction questionnaire at 6 months and 1 year

SECONDARY OUTCOMES:
Assessment of pain in patients receiving hypnosis sessions in cardiac surgery on the day of discharge from hospital, at 6 months and at 1 year. | 1 years
  Pain scale: EVS / EVA between 0 and 10
Assessment of stress and anxiety in patients receiving hypnosis at 6 months and 1 year. | 1 years
  EVA anxiety scale, satisfaction questionnaire between 0 and 10
Evaluation of quality of life at 6 months and 1 year. | 1 years
  EQ5D5L questionnaire on a scale between 0 and 100

CONTACTS AND LOCATIONS:
Locations (1):
- Delphine Rhem, Grenoble, France

IPD SHARING:
Plan to Share IPD: No
Analyses of the primary and secondary endpoints will be descriptive. Continuous variables will be described using the mean and standard deviation, as well as the median and interquartile range. Qualitative variables will be described in terms of numbers and associated percentages.
  All analyses will be carried out on a frozen database, in accordance with current good practice at Grenoble Alpes University Hospital.
  The analyses will be carried out under the supervision of a statistical engineer from the Data Engineering Unit.

REFERENCES:
- [Result] Ashton RC Jr, Whitworth GC, Seldomridge JA, Shapiro PA, Michler RE, Smith CR, Rose EA, Fisher S, Oz MC. The effects of self-hypnosis on quality of life following coronary artery bypass surgery: preliminary results of a prospective, randomized trial. J Altern Complement Med. 1995 Fall;1(3):285-90. doi: 10.1089/acm.1995.1.285. PMID 9395624
- [Result] de Klerk JE, du Plessis WF, Steyn HS, Botha M. Hypnotherapeutic ego strengthening with male South African coronary artery bypass patients. Am J Clin Hypn. 2004 Oct;47(2):79-92. doi: 10.1080/00029157.2004.10403627. PMID 15554461
- [Result] Schnur JB, Kafer I, Marcus C, Montgomery GH. HYPNOSIS TO MANAGE DISTRESS RELATED TO MEDICAL PROCEDURES: A META-ANALYSIS. Contemp Hypn. 2008 Aug 21;25(3-4):114-128. doi: 10.1002/ch.364. PMID 19746190
- [Result] Akgul A, Guner B, Cirak M, Celik D, Hergunsel O, Bedirhan S. The Beneficial Effect of Hypnosis in Elective Cardiac Surgery: A Preliminary Study. Thorac Cardiovasc Surg. 2016 Oct;64(7):581-588. doi: 10.1055/s-0036-1580623. Epub 2016 Apr 4. PMID 27043785
- [Result] Rousseaux F, Dardenne N, Massion PB, Ledoux D, Bicego A, Donneau AF, Faymonville ME, Nyssen AS, Vanhaudenhuyse A. Virtual reality and hypnosis for anxiety and pain management in intensive care units: A prospective randomised trial among cardiac surgery patients. Eur J Anaesthesiol. 2022 Jan 1;39(1):58-66. doi: 10.1097/EJA.0000000000001633. PMID 34783683
- [Result] Faymonville EM, Mambourg HP, Joris J, Vrijens B, Fissette J, Albert A, Lamy M. Psychological approaches during conscious sedation. Hypnosis versus stress reducing strategies: a prospective randomized study. Pain. 1997 Dec;73(3):361-367. doi: 10.1016/S0304-3959(97)00122-X. PMID 9469526
- [Result] Acikel MET. Evaluation of Depression and Anxiety in Coronary Artery Bypass Surgery Patients: A Prospective Clinical Study. Braz J Cardiovasc Surg. 2019 Aug 27;34(4):389-395. doi: 10.21470/1678-9741-2018-0426. PMID 31364347
- [Result] Ashton C Jr, Whitworth GC, Seldomridge JA, Shapiro PA, Weinberg AD, Michler RE, Smith CR, Rose EA, Fisher S, Oz MC. Self-hypnosis reduces anxiety following coronary artery bypass surgery. A prospective, randomized trial. J Cardiovasc Surg (Torino). 1997 Feb;38(1):69-75. PMID 9128126